CLINICAL TRIAL: NCT02280343
Title: OSCILLATION MECHANICS OF THE RESPIRATORY SYSTEM ASBESTOS EXPOSED : Early Diagnosis
Brief Title: Oscillation Mechanics of the Respiratory System Asbestos Exposed: Early Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Paula Morisco de Sá, OSCILLATION MECHANICS OF THE RESPIRATORY SYSTEM ASBESTOS EXPOSED : Early diagnosis, Rio de Janeiro State University
Other Study IDs: UERJ
Record Dates: First submitted 2014-10-24; First posted 2014-10-31 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Asbestosis
Keywords: forced oscillation tecnique; lung function; asbestosis
MeSH Terms: conditions — Asbestosis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: evaluated lung function — lung function tests

SUMMARY:
Inhalation of dust containing asbestos results in a process of interstitial pulmonary fibrosis called asbestosis. The Forced Oscillation Technique (FOT) evaluates the respiratory mechanics describing resistive, elastic and inertial properties. We believe that this technique may contribute to the early diagnosis of asbestosis.

DETAILED DESCRIPTION:
The aims of this study were (1) to use the FOT to analyze how respiratory mechanics is affected in patients with asbestos exposed, (2) to identify the best FOT parameters for the diagnosis of respiratory changes in these patients (3) Assess whether the presence of obstructive changes is associated with the smoking habit.The control group (CG) included 24 subjects with normal spirometric data and without a history of smoking or pulmonary disease formed by workers and students UERJ and FioCruz. Volunteers with asbestos exposure were from the Department of CESTEH/ FioCruz, totaling 24 exposed and 7 with diagnoses of asbestosis.

The diagnosis of asbestosis was established based on a history of substantial exposure to asbestos dusts and compatible radiological features, together with exclusion of other competing diagnoses.

The tests included a standardized questionnaire on respiratory symptoms, clinical evaluation; Plain radiography of the chest; FOT, plethysmography and spirometry, in that order.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of asbestosis

Exclusion Criteria:

* other diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: exposed to asbesto
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
changes in pulmonary mechanicals | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paula Sá, research, Principal Investigator — Universidade do Estado do Rio de Janeiro:Brazil
Locations (1):
- Paula Morisco de Sá, Rio de Janeiro, Rio de Janeiro, Brazil